CLINICAL TRIAL: NCT01300143
Title: Association of Conformational High-dose Radiotherapy and of Hyperselective Transarterial Chemoembolization in the Treatment of Hepatocellular Carcinoma
Acronym: TACERTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRD/10/06-M
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TACE (Active Comparator): Patients will be treated by 2 or 3 cures of hyperselective TACE. The first one at week 0 and the second one at week 8. If required, a third cure of TACE could be done at week16.
  Interventions: Other: TACE
- TACE + RTC (Experimental): Patients will be treated by one cure of TACE at week 0. Then, patients will be treated within two weeks by external conformational radiotherapy of 54 grey fractioned in 18 sessions during 3-4 weeks.
  Interventions: Other: TACE+ RTC

INTERVENTIONS:
Other: TACE — Control arm will be treated by 2 or 3 cures of TACE DC beads at week 0, 8 and 16 (if required)
  Arms: TACE
Other: TACE+ RTC — Experimental group will be treated by one cure of TACE DC Beads at week 0 then, within two weeks, by external conformational radiotherapy in 18 sessions
  Arms: TACE + RTC

SUMMARY:
Indication : Hepatocellular carcinoma, maximum size 9 cm, with single or multiple nodes whose total tumor mass can technically be irradiated, non-resectable, and not a candidate for percutaneous therapy with recommended treatment via hyperselective transarterial chemoembolisation (TACE).

DETAILED DESCRIPTION:
: Phase II controlled randomized trial, multicenter, comparing the benefit of additive conformational radiotherapy after therapy with hyperselective chemoembolisation (TACE) with treatment using three TACE treatments (standard of care).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age
* ECOG 0-1
* life expectancy ≥ 6 months
* Histologically proven hepatocellular carcinoma or proven according to radiological and biochemical criteria (EASL-AASLD) in cirrhotic patients
* Maximum lesion size ≤ 9 cm
* Non-eligible for surgery or percutaneous therapy
* Premature Child-Pugh A or B (7 points for the Child-Pugh score)
* AST and ALT < 7 x UNL
* Technical possibility of conformational external radiotherapy
* Technical possibility of TACE
* All the tumor mass must be able to be treated by TACE
* Written consent signed by the patient
* Patients affiliated to a social security system

Exclusion Criteria:

* Metastatic illness
* Minimal lesion size ≤ 5 mm
* Non controlled viral replication B
* History of radiotherapy at abdominal level
* Subjects capable of procreating without efficient contraception
* pregnancy or nursing female patient
* Contraindication of TACE or external conformational radiotherapy
* Any other concomitant experimental treatment
* Contraindication of Doxorubicin
* Patients who are unable to respect enslaving respiratory constraints if used by sites
* Patients who are unable to understand information and to follow protocol instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2018-10-26 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Time of tumor progression radiologically (CTScan) measured by mRECIST (Modified Response Evaluation Criteria In Solid Tumor). | up to 18 months

SECONDARY OUTCOMES:
Evaluation of the acute toxicity at the participants | within 90 days after the treatment
Evaluation of the late toxicity at the participants | after 90 days of treatment
Evaluation of the quality of life (assessed by QLQ-EORT C30) | the day of randomization (week 0), at week 12 and week 24
Evaluation of the rate of complete, partial response and stable disease after treatment (by RECIST criteria ) | at week 24,week 48 and week 72
Compare the health economic implications of these regimens in these patients. | up to18 months (week 72)
overall survival | within 3 years after first cure of TACE-DC BEADS

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille Feray, Pr, Principal Investigator — Henri Mondor Hospital (Paris)
Locations (18):
- France (18):
  - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - CH Avignon, Avignon
  - Institut Sainte Catherine, Avignon
  - CHU de Bordeaux, Bordeaux
  - AP-HP Henri Mondor, Créteil
  - CHU Dijon, Dijon
  - CHD les Oudairies, La Roche-sur-Yon
  - CHR de Lille Hôpital Claude Huriez, Lille
  - CHU de Lyon, Lyon
  - CHU de Nancy Hôpital Brabois, Nancy
  - CHU Nantes, Nantes
  - CHR Orléans, Orléans
  - AP-HP Paul Brousse Villejuif, Paris
  - Hôpital Tenon, Paris
  - La Pitié-Salpétrière, Paris
  - CHU de Reims, Reims
  - Centre Eugene Marquis, Rennes

REFERENCES:
- [Derived] Feray C, Campion L, Mathurin P, Archambreaud I, Mirabel X, Bronowicki JP, Rio E, Perret C, Mineur L, Oberti F, Touchefeu Y, Gournay J, Regnault H, Edeline J, Rode A, Hillion P, Blanc JF, Khac EN, Azoulay D, Luciani A, Preglisasco AG, Faurel-Paul E, Auble H, Mornex F, Merle P. TACE and conformal radiotherapy vs. TACE alone for hepatocellular carcinoma: A randomised controlled trial. JHEP Rep. 2023 Jan 29;5(4):100689. doi: 10.1016/j.jhepr.2023.100689. eCollection 2023 Apr. PMID 36937990